CLINICAL TRIAL: NCT00612586
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Study of Enzastaurin With 5-FU/LV Plus Bevacizumab as Maintenance Regimen Following First Line Therapy for Metastatic Colorectal Cancer
Brief Title: Study of Enzastaurin With 5-Fluorouracil/Leucovorin (5-FU/LV) Plus Bevacizumab as Maintenance Regimen Following First Line Therapy for Metastatic Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10534; H6Q-MC-S064 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — enzastaurin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzastaurin + 5-FU/LV + Bev (Experimental): 5-fluorouracil/leucovorin (5-FU/LV) plus bevacizumab (Bev) in combination with enzastaurin
  Interventions: Drug: Enzastaurin; Drug: Leucovorin (LV); Drug: 5-fluorouracil (5-FU); Drug: Bevacizumab (Bev)
- Placebo + 5-FU/LV + Bev (Placebo Comparator): 5-fluorouracil/leucovorin (5-FU/LV) plus bevacizumab (Bev) in combination with placebo
  Interventions: Drug: Placebo; Drug: Leucovorin (LV); Drug: 5-fluorouracil (5-FU); Drug: Bevacizumab (Bev)

INTERVENTIONS:
Drug: Enzastaurin — 1125 milligram (mg) loading dose, then 250 mg twice daily, oral up to 1 year (yr) or until progressive disease
  Other Names: LY317615
  Arms: Enzastaurin + 5-FU/LV + Bev
Drug: Placebo — oral, daily (up to 1 yr or until progressive disease)
  Arms: Placebo + 5-FU/LV + Bev
Drug: Leucovorin (LV) — 400 milligram per meter squared (mg/m^2) intravenously (IV), Day 1 of 14 day cycle (up to 1 yr or until progressive disease)
Drug: 5-fluorouracil (5-FU) — 400 mg/m^2 bolus then 2400 mg/m^2 IV over 46 hours, Day 1 of 14 day cycle (up to 1 yr or until progressive disease)
Drug: Bevacizumab (Bev) — 5 milligram per kilogram (mg/kg) IV, Day 1 of 14 day cycle (up to 1 yr or until progressive disease)

SUMMARY:
This study will evaluate the addition of enzastaurin to 5-FU (5-fluorouracil)/LV (leucovorin) plus bevacizumab in the maintenance of best response obtained with 6 cycles of first-line therapy consisting of 5-FU/LV + oxaliplatin (FOLFOX) or 5-FU/LV + irinotecan (FOLFIRI), plus bevacizumab in patients with Metastatic Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of locally advanced or metastatic colorectal cancer (CRC) that is not curable. The histology types to be included are adenocarcinoma, mucinous adenocarcinoma, signet ring, and undifferentiated. Patients with neuroendocrine carcinomas will be excluded.
* Received 6 cycles (3 months [12 weeks]) of first-line therapy with FOLFOX or FOLFIRI, plus bevacizumab for metastatic CRC. Patients have received at least 5 cycles with bevacizumab. Patients who received 6 cycles of first-line therapy with FOLFOX or FOLFIRI, plus bevacizumab for recurrent CRC that has relapsed at least 12 months after completion of adjuvant therapy will also be included. All standard FOLFOX (FOLFIRI) regimens given on a biweekly schedule will be permitted; however, 21-day regimens will not be allowed.
* No more than 4 weeks may pass between the end of first-line therapy (that is, Day 14 of Cycle 6) and randomization.
* Documented evidence of tumor response of complete response (CR), partial response (PR), or stable disease (SD) by computed tomography (CT) scan or magnetic resonance imaging (MRI). Confirmation of response is not required.

Exclusion Criteria:

* Are unable to swallow tablets.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have known central nervous system metastases.
* Are receiving concurrent administration of any other antitumor therapy.
* Patients who have significant heart, liver, kidney, or psychiatric disease or have an active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krems
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clichy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Weiden
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico

REFERENCES:
- [Derived] Wolff RA, Fuchs M, Di Bartolomeo M, Hossain AM, Stoffregen C, Nicol S, Heinemann V. A double-blind, randomized, placebo-controlled, phase 2 study of maintenance enzastaurin with 5-fluorouracil/leucovorin plus bevacizumab after first-line therapy for metastatic colorectal cancer. Cancer. 2012 Sep 1;118(17):4132-8. doi: 10.1002/cncr.26692. Epub 2011 Dec 27. PMID 22213153
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzastaurin + 5-FU/LV + Bev: Enzastaurin: Loading dose of 1125 milligrams (mg) orally, 3 times during Day 1 of Cycle 1 (14-day cycle); 500 mg orally, twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  Leucovorin (LV): 400 mg per meter squared (mg/m^2) intravenously (IV) on Day 1 of each 14-day cycle, followed by 5-fluorouracil (5-FU) 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bevacizumab (Bev): 5 milligrams/kilogram (mg/kg) IV.
  First-line therapy for metastatic colorectal cancer (CRC) received prior to entering the study: six 14-day cycles (12 weeks) folinic acid, 5-FU, and oxaliplatin (FOLFOX) or folinic acid, 5-FU, and irinotecan (FOLFIRI), plus Bev.
- Placebo + 5-FU/LV + Bev: Placebo: Orally 3 times during Day 1 of Cycle 1 (14-day cycle); orally, twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  LV: 400 mg/m^2 IV on Day 1 of each 14-day cycle, followed by 5-FU 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bev: 5 mg/kg IV.
  First-line therapy for CRC received prior to entering the study: six 14-day cycles (12 weeks) FOLFOX or FOLFIRI, plus Bev.
Period: Overall Study
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5-FU/LV + Bev
Started | 58 | 59
Received at Least 1 Dose | 57 | 58
Completed | 15 | 18
Not Completed | 43 | 41
Not completed — Adverse Event | 6 | 2
Not completed — Death | 1 | 0
Not completed — Entry Criteria Not Met | 0 | 2
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Physician Decision | 1 | 2
Not completed — Sponsor Decision | 1 | 1
Not completed — Progressive Disease | 26 | 24
Not completed — Randomized and Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Enzastaurin + 5-FU/LV + Bev: Enzastaurin: Loading dose of 1125 mg orally, 3 times during Day 1 of Cycle 1 (14-day cycle); 500 mg orally, twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  LV: 400 mg/m^2 IV on Day 1 of each 14-day cycle, followed by 5-FU 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bev: 5 mg/kg IV.
  First-line therapy for metastatic CRC received prior to entering the study: six 14-day cycles (12 weeks) folinic acid, 5-FU, and oxaliplatin (FOLFOX) or folinic acid, 5-FU, and irinotecan (FOLFIRI), plus Bev.
- Placebo + 5-FU/LV + Bev: Placebo: administered orally 3 times during Day 1 of Cycle 1 (14 day cycle); placebo administered orally twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  Leucovorin (LV): 400 mg/m^2 administered by IV on Day 1 of each 14 day cycle, followed by 5-fluorouracil (5-FU) 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bevacizumab (Bev): 5 milligrams/kilogram (mg/kg) IV.
  First-line therapy for CRC received prior to entering the study: six 14-day cycles (12 weeks) folinic acid, 5-fluorouracil (5-FU), and oxaliplatin (FOLFOX) or folinic acid, 5-FU, and irinotecan (FOLFIRI), plus Bev.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5-FU/LV + Bev | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.55 (10.90) | 62.49 (9.48) | 62.52 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 37 | 38 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 55 | 54 | 109
  African | 1 | 2 | 3
  Hispanic | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 5 | 8 | 13
  France | 6 | 3 | 9
  Germany | 12 | 17 | 29
  Italy | 13 | 16 | 29
  United States | 22 | 15 | 37
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG a scale to rate participants' activity status: 0-fully active; 1-Ambulatory, Restricted Strenuous Activity; 2-Ambulatory, No Work Activities; 3-Partially Confined to Bed, Limited Self Care; 4-Completely Disabled.
  Participants
    0 | 42 | 45 | 87
    1 | 16 | 13 | 29
    2 | 0 | 1 | 1
Initial Pathological Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma, Mucinous, Not Otherwise Specified | 3 | 4 | 7
  Adenocarcinoma, Colon | 55 | 54 | 109
  Unknown or Not Reported | 0 | 1 | 1
Stage of Disease at Study Entry [Count of Participants; unit: Participants] — Tumor Stage (St) I-in inner lining or muscle layer of bowel wall; St IIa-in outer layer of bowel wall or invades adjacent tissues; St IIb- invaded adjacent organs or penetrates peritoneum; St IIIa- in inner lining or muscle layer of bowel wall and has spread to 1-3 nearby nodes; St IIIb- in outer layer of bowel wall or invades adjacent tissue or organs, and has spread to 1-3 nearby nodes; St IIIc-in outer layer of bowel wall or invades adjacent tissue or organs, and has spread to ≥ 4 nearby nodes; St IV- has spread to distant sites. Tumor stage is missing for some participants.
  Participants
    I | 0 | 0 | 0
    IIa | 0 | 1 | 1
    IIb | 0 | 0 | 0
    IIIa | 0 | 0 | 0
    IIIb | 4 | 0 | 4
    IIIc | 2 | 1 | 3
    IV | 47 | 52 | 99
    Unknown or Not Reported | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first observation of disease progression or death due to any cause. Progressive disease was determined using a modified version of Response Evaluation Criteria in Solid Tumor (RECIST) Assessment and was defined as at least a 20% increase in sum of longest diameter of target lesions. Time to disease progression was censored at the date of death if death was due to other cause.
Time Frame: Randomization to measured progressive disease or death up to 17.2 months
Population: Intent-to-Treat (ITT) Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Placebo + 5FU/LV + Bev: Placebo: Orally 3 times during Day 1 of Cycle 1 (14-day cycle); orally, twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  LV: 400 mg/m^2 IV on Day 1 of each 14-day cycle, followed by 5-FU 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bev: 5 mg/kg IV.
  First-line therapy for CRC received prior to entering the study: six 14-day cycles (12 weeks) FOLFOX or FOLFIRI, plus Bev.
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5FU/LV + Bev
Number analyzed (Participants) | 58 | 59
months | 5.8 [4.4 to 7.8] | 8.1 [6.8 to 12.1]
Statistical Analysis 1: Comparison: Enzastaurin + 5-FU/LV + Bev vs Placebo + 5FU/LV + Bev; Test type: Superiority or Other; p = 0.8956, Log Rank — One sided

2. Secondary Outcome: Overall Survival (OS)
Description: OS was the duration from enrollment to death due to any cause. For participants who are alive, OS is censored at the last contact.
Time Frame: Randomization up to 22.8 months
Population: ITT Population: All randomized participants; Number of participants censored was 54 in Placebo + 5-FU/LV + Bev treatment group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5FU/LV + Bev
Number analyzed (Participants) | 58 | 59
months | NA [13.1 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [15.3 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Enzastaurin + 5-FU/LV + Bev vs Placebo + 5FU/LV + Bev; Test type: Superiority or Other; p = 0.9865, Log Rank — One-sided

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A summary of serious and all other non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Randomization up to 17.2 months
Population: Safety Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + 5FU/LV +Bev: Placebo: Orally 3 times during Day 1 of Cycle 1 (14-day cycle); orally, twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  LV: 400 mg/m^2 IV on Day 1 of each 14-day cycle, followed by 5-FU 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bev: 5 mg/kg IV.
  First-line therapy for CRC received prior to entering the study: six 14-day cycles (12 weeks) FOLFOX or FOLFIRI, plus Bev.
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5FU/LV +Bev
Number analyzed (Participants) | 57 | 58
Participants
  Serious AEs | 15 | 11
  Other Non-Serious AEs | 53 | 52

4. Secondary Outcome: Overall Survival (OS) From Start of First Line Therapy
Description: OS was the duration from first line therapy to death due to any cause. For participants who are alive, OS is censored at the last contact.
Time Frame: Start of first line therapy (approximately 3 months prior to randomization) to date of death from any cause up to 27 months post randomization
Population: ITT Population: All randomized participants; Number of participants censored were 45 in Enzastaurin + 5-FU/LV + Bev treatment group and 54 in Placebo + 5-FU/LV + Bev treatment group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5FU/LV + Bev
Number analyzed (Participants) | 58 | 59
months | 20.0 [15.6 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [19.0 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment.

5. Secondary Outcome: PFS From Start of First Line Therapy
Description: PFS was defined as the time from first line therapy to the first observation of disease progression or death due to any cause. Progressive disease was determined using a modified version of RECIST Assessment and was defined as at least a 20% increase in sum of longest diameter of target lesions. Time to disease progression was censored at the date of death if death was due to other cause.
Time Frame: Start of first line therapy to measured progressive disease or death up to 24 months
Population: ITT Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin + 5-FU/LV + Bev | Placebo + 5FU/LV + Bev
Number analyzed (Participants) | 58 | 59
months | 8.9 [7.5 to 11.0] | 11.3 [10.3 to 15.6]

ADVERSE EVENTS:
Groups:
- Enzastaurin + 5-FU/LV Plus Bevacizumab: Enzastaurin: loading dose of 1125 mg administered orally 3 times during Day 1 of Cycle 1 (14 day cycle); 500 mg administered orally twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  Leucovorin (LV): 400 mg per meter squared (mg/m^2) administered by IV on Day 1 of each 14 day cycle, followed by 5-fluorouracil (5-FU) 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bevacizumab (Bev): 5 milligrams/kilogram (mg/kg) IV.
  First-line therapy for CRC received prior to entering the study: six 14-day cycles (12 weeks) folinic acid, 5-fluorouracil (5-FU), and oxaliplatin (FOLFOX) or folinic acid, 5-FU, and irinotecan (FOLFIRI), plus Bev.
- Placebo + 5FU/LV + Bevacizumab: Placebo: administered orally 3 times during Day 1 of Cycle 1 (14 day cycle); placebo administered orally twice daily on Day 2 to Day 14 of Cycle 1 and all subsequent cycles.
  Leucovorin (LV): 400 mg/m^2 administered by IV on Day 1 of each 14 day cycle, followed by 5-fluorouracil (5-FU) 400 mg/m^2 IV bolus then 2400 mg/m^2 IV over 46 hours, plus Bevacizumab (Bev): 5 milligrams/kilogram (mg/kg) IV.
  First-line therapy for CRC received prior to entering the study: six 14-day cycles (12 weeks) folinic acid, 5-fluorouracil (5-FU), and oxaliplatin (FOLFOX) or folinic acid, 5-FU, and irinotecan (FOLFIRI), plus Bev.
Arm/Group | Enzastaurin + 5-FU/LV Plus Bevacizumab | Placebo + 5FU/LV + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 15/57 | 11/58
Other Adverse Events (participants affected / at risk) | 53/57 | 52/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin + 5-FU/LV Plus Bevacizumab (N=57) | Placebo + 5FU/LV + Bevacizumab (N=58)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Stent malapposition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin + 5-FU/LV Plus Bevacizumab (N=57) | Placebo + 5FU/LV + Bevacizumab (N=58)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (14) | 7 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (11) | 8 (12)
Eye irritation (Eye disorders) | 2 (2) | 3 (3)
Lacrimation increased (Eye disorders) | 3 (3) | 3 (3)
Vision blurred (Eye disorders) | 3 (3) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 5 (6)
Constipation (Gastrointestinal disorders) | 13 (15) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 19 (25) | 22 (33)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 5 (5) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (6) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (18) | 15 (27)
Oral pain (Gastrointestinal disorders) | 5 (6) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7) | 10 (15)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 24 (29) | 23 (29)
Mucosal inflammation (General disorders) | 9 (12) | 9 (12)
Pain (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 7 (8)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (3)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (5) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (5)
Blood creatinine increased (Investigations) | 2 (2) | 3 (3)
Haemoglobin decreased (Investigations) | 6 (6) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3) | 2 (2)
Urine colour abnormal (Investigations) | 7 (7) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 6 (11)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 10 (17) | 8 (12)
Neuropathy peripheral (Nervous system disorders) | 4 (5) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (5) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (7) | 8 (8)
Polyneuropathy (Nervous system disorders) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 4 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Chromaturia (Renal and urinary disorders) | 4 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (6) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 13 (16)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (16) | 14 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 5 (5)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 7 (7) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days